CLINICAL TRIAL: NCT06678828
Title: Establishing the Clinical Utility of ClarityDX Prostate
Brief Title: Clinical Utility of ClarityDX Prostate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanostics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: APCaRI-08
Record Dates: First submitted 2024-09-26; First posted 2024-11-07 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: ClarityDX Prostate; Utility Study; Clinical Utility of ClarityDX Prostate; Establishing the Clinical Utility of ClarityDX Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control (Other): Control/Standard of Care arm- ClarityDX Prostate will be run for these participants. Participants and healthcare providers will be blinded to the results report and participants will be considered for prostate MRI/advanced imaging and /or biopsy based on standard clinical criteria. The results of the ClarityDX Prostate will be unblinded to the study teams at the 12 months follow-up visit. The study team will then share the test results with the participant's health care team to assess whether there is a need to change the participant's care path.
  Interventions: Other: ClarityDX Prostate, blinded
- ClarityDX Prostate (Experimental): The report will be shared with the healthcare team of participants randomized into the ClarityDX Prostate arm before the healthcare team decides whether to perform an MRI/advanced imaging and/or biopsy.
  Interventions: Other: ClarityDX Prostate

INTERVENTIONS:
Other: ClarityDX Prostate — The ClarityDX Prostate report will be shared with the healthcare team of participants randomized into ClarityDX Prostate arm before the healthcare team decides whether to perform an MRI/advanced imaging and/or biopsy.
  Arms: ClarityDX Prostate
Other: ClarityDX Prostate, blinded — ClarityDX Prostate will be run for the control participants. Participants (and healthcare team) in the control arm will be blinded to the ClarityDX Prostate results and will be considered for prostate MRI/advanced imaging and/or biopsy based on standard of care criteria. The result of the ClarityDX Prostate will be unblinded to study teams at the 12 months follow-up visit (± 2 months). The study team will then share the test results with the participant's health care team to assess whether there is a need to change the participant's care path.
  Arms: The control

SUMMARY:
ClarityDX Prostate builds upon the utility of total and free PSA as well as simple clinical features in a decision support model to determine a patient's risk of having clinically significant prostate cancer. The highly accurate ClarityDX Prostate risk score enables clinicians and patients to collectively make more informed decisions regarding the appropriateness of subsequent imaging or biopsy procedures. The clinical pathway aligns with the Canadian Urological Association (CUA) to use adjunctive strategies to better stratify risk of clinically significant prostate cancer.

ClarityDX Prostate consists of four separate models that can be used depending on the information available:

1. ClarityDX Prostate. This model incorporates the patient's total PSA and free PSA levels as well as the age of the patient and whether they have had a previous negative biopsy.
2. ClarityDX Prostate + DRE. This model incorporates ClarityDX Prostate + DRE (normal or abnormal DRE findings).
3. ClarityDX Prostate + MRI. This model incorporates ClarityDX Prostate + MRI (PI-RADS score and prostate volume as determined from an mpMRI scan).
4. ClarityDX Prostate + MRI + DRE. This model incorporates ClarityDX Prostate + MRI + DRE.

PRIMARY OBJECTIVE The purpose of this study is to investigate the clinical utility of ClarityDX Prostate on in reducing further healthcare utilization for men identified to be at risk of prostate cancer.

SECONDARY OBJECTIVES

* Assess the effect of ClarityDX Prostate on the proportion of negative biopsies and biopsies diagnosing Gleason Grade (GG)<2.
* Measure the difference in MRI numbers between the test and control groups.
* Evaluate the effect of ClarityDX Prostate on the prioritization of healthcare services to participants with high-risk of having clinically significant prostate cancer.
* Infer the potential to use ClarityDX Prostate for prostate cancer screening to inform urology referral.
* Perform a health economics assessment and cost-benefit analysis for the use of ClarityDX Prostate.

This is a prospective, randomized, two-armed clinical utility study that will enroll participants referred to urology clinics for suspicion of prostate cancer. The arms of the study are ClarityDX Prostate and Standard of Care (SOC).

DETAILED DESCRIPTION:
When stratifying patients for prostate cancer, it is ideal to avoid delay in treating high-risk participants that do require a biopsy, while avoiding unnecessary procedures in low-risk patients. The purpose of this study is to investigate in a real-world setting whether the use of ClarityDX Prostate would further reduce potentially unnecessary healthcare utilization of men referred to urology clinics with suspicion of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years of age
2. Referred to urology for suspicion of prostate cancer
3. No prior prostate cancer diagnosis
4. Willing to participate in the study
5. Availability for cancer care in the jurisdiction of recruitment

Exclusion Criteria:

1. Unwilling to participate in the study
2. Unable to consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1074 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who receive biopsy and are not diagnosed with clinically significant prostate cancer | 12 months
  'Not diagnosed with clinically significant prostate cancer' refers to biopsies that show no cancer or clinically insignificant cancer

SECONDARY OUTCOMES:
Proportion of patients diagnosed with clinically significant prostate cancer | 12 months
Proportion of patients who undergo advanced imaging | 12 months
Proportion of patients who undergo biopsy | 12 months
Time from first urologist consultation to clinically significant prostate cancer diagnosis | 12 months
  Time in days from seeing urologist for the first time to getting diagnosed with cancer
Number of biopsies deferred | 12 months
  A biopsy deferred is a biopsy that was ordered by the physicians but was not performed
Inferred usability of ClarityDX Prostate for prostate cancer screening prior to urology referral | 12 months
Inferred reduction in referrals to urology by family physicians as a result of a low-Risk Score from ClarityDX Prostate | 12 months
Comparison of associated healthcare costs with and without the use of ClarityDX Prostate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam Kinnaird, MD PhD FRCSC, Principal Investigator — University of Alberta; M Eric Hyndman, MD, PhD, FRCSC, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Prostate Cancer Centre, Calgary, Alberta
  - Kipnes Urology Centre, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hyndman ME, Paproski RJ, Kinnaird A, Fairey A, Marks L, Pavlovich CP, Fletcher SA, Zachoval R, Adamcova V, Stejskal J, Aprikian A, Wallis CJD, Pink D, Vasquez C, Beatty PH, Lewis JD. Development of an effective predictive screening tool for prostate cancer using the ClarityDX machine learning platform. NPJ Digit Med. 2024 Jun 20;7(1):163. doi: 10.1038/s41746-024-01167-9. PMID 38902526
- See also: Related Info — https://www.nanosticsdx.com/
- See also: Related Info — https://apcari.ca/